CLINICAL TRIAL: NCT01818427
Title: Prehospital Air Medical Plasma (PAMPer) Phase III Multicenter, Prospective, Randomized, Open-label, Interventional Trial A Four Year Multicenter Open Label Randomized Trial
Brief Title: PreHospital Air Medical Plasma Trial
Acronym: PAMPer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jason Sperry (Other)
Collaborators: University of Texas (Other); University of Louisville (Other); Vanderbilt University (Other); Case Western Reserve University (Other); The University of Tennessee, Knoxville (Other); JPS Health Network (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Jason Sperry, MD, MPH, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11152002 IND 15117
Record Dates: First submitted 2013-03-19; First posted 2013-03-26 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Hemmorhagic Shock During Air Medical Transport
Keywords: hemmorhagic shock, plasma, air medical transport, randomized, multicenter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- plasma (Experimental): infusion of 2 units of plasma
  Interventions: Biological: infusion of 2 units of plasma
- standard air medical care (No Intervention): control group

INTERVENTIONS:
Biological: infusion of 2 units of plasma — infusion of 2 units of plasma
  Arms: plasma

SUMMARY:
To determine the effect of the prehospital infusion during air transport of 2 units of AB plasma on 30 day mortality in patients with hemorrhagic shock as compared to conventional care.

DETAILED DESCRIPTION:
Background: Although advances in the care of the severely injured patient have occurred over the last decade, patients continue to be plagued with uncontrolled hemorrhage resulting in significant early mortality and the development of multiple organ failure and associated complications. A primary driving force for this unbridled hemorrhage has been shown to be the early coagulopathy which complicates severe injury. Increasing evidence suggests that blood component transfusion protocols that address this early coagulopathy, once a patient arrives at a trauma center, are associated with lower mortality and a reduction in blood component transfusion requirements. Prehospital interventions which quell this early coagulopathy in an earlier setting have the potential to minimize or even prevent this vicious hemorrhagic cascade, further lowering blood component transfusion requirements and reducing the resultant morbid sequelae which complicates severe injury.

Objective/Hypothesis: The primary hypothesis will be that prehospital infusion of plasma during air medical transport in patients with hemorrhagic shock will lower 30 day mortality. The secondary hypotheses include that prehospital infusion of plasma will reduce 24 hour blood transfusion, multiple organ failure, nosocomial infection, and acute lung injury, reduce or prevent the early coagulopathy as demonstrated by improving presenting coagulation and thromboelastography parameters, and reduce the early inflammatory cytokine response, thrombomodulin and increase protein C levels.

ELIGIBILITY:
Inclusion Criteria: Hemorrhagic shock not responsive to crystalloid infusion -

Exclusion Criteria: Isolated Fall, Cervical cord injury, prisoner, pregnant patient, traumatic arrest

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2014-05; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Sperry, MD,MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Lorence JM, Donohue JK, Iyanna N, Guyette FX, Gimbel E, Brown JB, Daley BJ, Eastridge BJ, Miller RS, Nirula R, Harbrecht BG, Claridge JA, Phelan HA, Vercruysse G, O'Keeffe T, Joseph B, Neal MD, Sperry JL. Characterization of adverse events in injured patients at risk of hemorrhagic shock: a secondary analysis of three harmonized prehospital randomized clinical trials. Trauma Surg Acute Care Open. 2024 Jun 25;9(1):e001465. doi: 10.1136/tsaco-2024-001465. eCollection 2024. PMID 38933603
- [Derived] Wu J, Moheimani H, Li S, Kar UK, Bonaroti J, Miller RS, Daley BJ, Harbrecht BG, Claridge JA, Gruen DS, Phelan HA, Guyette FX, Neal MD, Das J, Sperry JL, Billiar TR. High Dimensional Multiomics Reveals Unique Characteristics of Early Plasma Administration in Polytrauma Patients With TBI. Ann Surg. 2022 Oct 1;276(4):673-683. doi: 10.1097/SLA.0000000000005610. Epub 2022 Jul 19. PMID 35861072
- [Derived] Gruen DS, Guyette FX, Brown JB, Okonkwo DO, Puccio AM, Campwala IK, Tessmer MT, Daley BJ, Miller RS, Harbrecht BG, Claridge JA, Phelan HA, Neal MD, Zuckerbraun BS, Yazer MH, Billiar TR, Sperry JL. Association of Prehospital Plasma With Survival in Patients With Traumatic Brain Injury: A Secondary Analysis of the PAMPer Cluster Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2016869. doi: 10.1001/jamanetworkopen.2020.16869. PMID 33057642
- [Derived] Gruen DS, Brown JB, Guyette FX, Vodovotz Y, Johansson PI, Stensballe J, Barclay DA, Yin J, Daley BJ, Miller RS, Harbrecht BG, Claridge JA, Phelan HA, Neal MD, Zuckerbraun BS, Billiar TR, Sperry JL; PAMPer study group. Prehospital plasma is associated with distinct biomarker expression following injury. JCI Insight. 2020 Apr 23;5(8):e135350. doi: 10.1172/jci.insight.135350. PMID 32229722
- [Derived] Pusateri AE, Moore EE, Moore HB, Le TD, Guyette FX, Chapman MP, Sauaia A, Ghasabyan A, Chandler J, McVaney K, Brown JB, Daley BJ, Miller RS, Harbrecht BG, Claridge JA, Phelan HA, Witham WR, Putnam AT, Sperry JL. Association of Prehospital Plasma Transfusion With Survival in Trauma Patients With Hemorrhagic Shock When Transport Times Are Longer Than 20 Minutes: A Post Hoc Analysis of the PAMPer and COMBAT Clinical Trials. JAMA Surg. 2020 Feb 1;155(2):e195085. doi: 10.1001/jamasurg.2019.5085. Epub 2020 Feb 19. PMID 31851290
- [Derived] Sperry JL, Guyette FX, Brown JB, Yazer MH, Triulzi DJ, Early-Young BJ, Adams PW, Daley BJ, Miller RS, Harbrecht BG, Claridge JA, Phelan HA, Witham WR, Putnam AT, Duane TM, Alarcon LH, Callaway CW, Zuckerbraun BS, Neal MD, Rosengart MR, Forsythe RM, Billiar TR, Yealy DM, Peitzman AB, Zenati MS; PAMPer Study Group. Prehospital Plasma during Air Medical Transport in Trauma Patients at Risk for Hemorrhagic Shock. N Engl J Med. 2018 Jul 26;379(4):315-326. doi: 10.1056/NEJMoa1802345. PMID 30044935
- [Derived] Reynolds PS, Michael MJ, Cochran ED, Wegelin JA, Spiess BD. Prehospital use of plasma in traumatic hemorrhage (The PUPTH Trial): study protocol for a randomised controlled trial. Trials. 2015 Jul 30;16:321. doi: 10.1186/s13063-015-0844-5. PMID 26220293

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plasma | Standard Air Medical Care
Started | 239 | 284
Completed | 230 | 271
Not Completed | 9 | 13

BASELINE CHARACTERISTICS:
Population: 22 patients total, 8 in the plasma arm and 12 in the standard care arm withdrew consent and 1 patient in each arm was a prisoner and could not be included in the analysis cohort
Groups:
- Total: Total of all reporting groups
Arm/Group | Plasma | Standard Air Medical Care | Total
Number analyzed (Participants) | 230 | 271 | 501
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [31 to 59] | 46 [28 to 60] | 45 [29 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 71 | 137
  Male | 164 | 200 | 364
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 29 | 43
  White | 207 | 228 | 435
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 13 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 230 | 271 | 501

OUTCOME MEASURES:

1. Primary Outcome: Our Primary Outcome for the Proposal Will be 30 Day Mortality
Description: All cause 30 day mortality using imputation for those with missing 30 day mortality.
Time Frame: 30 days
Population: 10 patients in each arm were lost to follow-up for 30-day mortality and 22 patients total, 8 in the plasma arm and 12 in the standard care arm withdrew consent and 1 patient in each arm was a prisoner and could not be included in the analysis cohort. We compared 30-day mortality using a two sided pooled z test with continuity correction.
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard Air Medical Care
Number analyzed (Participants) | 220 | 261
Participants | 53 | 89

2. Secondary Outcome: Twenty Four-Hour Blood Transfusion Requirements
Description: 24-hour blood transfusion requirements will be determined by recording blood volume (mls) and number of Units transfused from the time of trauma bay arrival or upon completion of pre-hospital initiated plasma infusion. For survival bias analysis, volumes and number of blood transfusion Units received at 3, 6, 12, and 18 hours will also be recorded.
Time Frame: at twenty four hours
Measure: Median (Inter-Quartile Range); unit: units of blood
Arm/Group | Plasma | Standard Air Medical Care
Number analyzed (Participants) | 230 | 271
units of blood | 3 [0 to 7] | 4 [1 to 9]

3. Secondary Outcome: In-hospital Mortality
Description: In hospital mortality will be prospectively recorded from the time of trauma bay arrival. Over the first 24 hours we will document and record the time of death in hours, while after the 24 hour time point, we will document and record the time of death in days from arrival. We suspect that patients in hemorrhagic shock will have a significant percentage of mortality occurring in the first 24 hour period.
Time Frame: during hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard Air Medical Care
Number analyzed (Participants) | 230 | 271
Participants | 51 | 88

4. Secondary Outcome: Multiple Organ Failure
Description: Organ dysfunction will be evaluated via a well-validated scoring system referred to as the Multiple Organ Dysfunction Score (MODScore). Patients who are never admitted to the ICU or those with a length of ICU stay of less than 48 hours will be considered to have a MODScore of 0. A summary of the MODScore may be calculated by summing the worst scores of each of the individual systems over the course of the ICU stay (Table 1). A summary MODScore > 5 will be classified as multiple organ failure (MOF). Scores will be determined daily up until post injury day 28 or ICU discharge.
Time Frame: during hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard Air Medical Care
Number analyzed (Participants) | 230 | 271
Participants | 145 | 156

5. Secondary Outcome: Acute Lung Injury (ALI) and Transfusion Related Acute Lung Injury (TRALI)
Description: Development of ALI will be assessed which includes: 1) bilateral infiltrates on chest x-ray, 2) a capillary wedge pressure < 18mmHg, and 3) Pao2/Fio2 ratio < 300 via blood gas analysis. In those patients without a Swan-Ganz catheter to determine capillary wedge pressure, the absence of signs of, or clinical concern, for elevated left sided atrial pressures will be used for the diagnosis. All patients who remain intubated beyond the first 24 hours post-injury will be evaluated using blood gas analysis and chest x-ray evaluation. Those patients who remain intubated at 48 hours through 7 days will be reevaluated for this outcome at these time points. The diagnosis of TRALI will be defined as when ALI occurs within the first 6 hours from arrival at the trauma center as it is clinically defined.
Time Frame: hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Plasma | Standard Air Medical Care
Number analyzed (Participants) | 230 | 271
Participants | 48 | 50

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Plasma | Standard Air Medical Care
All-Cause Mortality (participants affected / at risk) | 53/220 | 89/261
Serious Adverse Events (participants affected / at risk) | 1/220 | 2/261
Other Adverse Events (participants affected / at risk) | 5/220 | 2/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plasma (N=220) | Standard Air Medical Care (N=261)
tranfusion-related reaction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
adult respirator distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plasma (N=220) | Standard Air Medical Care (N=261)
allergic reation (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaphylaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
fever (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
hypotension (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
urticaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT01818427/Prot_SAP_000.pdf